CLINICAL TRIAL: NCT03114657
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Study of Crenezumab in Patients With Prodromal to Mild Alzheimer's Disease
Brief Title: A Study of Crenezumab Versus Placebo to Evaluate the Efficacy and Safety in Participants With Prodromal to Mild Alzheimer's Disease (AD)
Acronym: CREAD 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was discontinued due to an interim analysis in the BN29552 study, which indicated that Crenezumab was unlikely to meet its primary endpoint.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN29553; 2016-003288-20 (EudraCT Number)
Record Dates: First submitted 2017-03-28; First posted 2017-04-14 (Actual); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received intravenous (IV) infusion of Placebo every 4 weeks (Q4W) for 100 weeks.
  Interventions: Drug: Placebo
- Crenezumab (Experimental): Participants received intravenous (IV) infusion of Crenezumab every 4 weeks (Q4W) for 100 weeks.
  Interventions: Drug: Crenezumab

INTERVENTIONS:
Drug: Crenezumab — Crenezumab was administered by intravenous (IV) infusion at 60mg/kg as per the dosing schedule described above.
  Arms: Crenezumab
Drug: Placebo — Placebo was administered by intravenous (IV) infusion at 60mg/kg as per the dosing schedule described above.
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel-group study will evaluate the efficacy and safety of crenezumab versus placebo in participants with prodromal to mild AD. Participants will be randomized 1:1 to receive either intravenous (IV) infusion of crenezumab or placebo every 4 weeks (Q4W) for 100 weeks. The primary efficacy assessment will be performed at 105 weeks. The participants who do not enter open-label extension will enter for a long term follow-up period for up to 52 weeks after the last crenezumab dose (Week 153).

ELIGIBILITY:
Inclusion Criteria:

* Weight between 40 and 120 kilograms (Kg) inclusive
* Availability of a person (referred to as the "caregiver") who in the investigator's judgment:
* Has frequent and sufficient contact with the participant to be able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits (which require partner input for scale completion), signs the necessary consent form, and has sufficient cognitive capacity to accurately report upon the participant's behavior and cognitive and functional abilities
* Fluency in the language of the tests used at the study site
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing (eye glasses and hearing aids are permitted)
* Evidence of the AD pathological process, by a positive amyloid assessment either on cerebrospinal fluid (CSF) amyloid beta 1-42 levels as measured on the Elecsys beta-amyloid(1-42) test system or amyloid PET scan by qualitative read by the core/central PET laboratory
* Demonstrated abnormal memory function at screening (up to 4 weeks before screening begins) or screening (FCSRT cueing index =<0.67 AND free recall =<27)
* Screening mini mental state examination (MMSE) score of greater than or equal to (>=) 22 points and Clinical Dementia Rating-Global Score (CDR-GS) of 0.5 or 1.0
* Meets National Institute on Aging/Alzheimer's Association (NIAAA) core clinical criteria for probable AD dementia or prodromal AD (consistent with the NIAAA diagnostic criteria and guidelines for mild cognitive impairment (MCI)
* If receiving symptomatic AD medications, the dosing regimen must have been stable for 3 months prior to screening
* Participant must have completed at least 6 years of formal education after the age of 5 years

Exclusion Criteria:

* Any evidence of a condition other than AD that may affect cognition such as other dementias, stroke, brain damage, autoimmune disorders (e.g. multiple sclerosis) or infections with neurological sequelae.
* History of major psychiatric illness such as schizophrenia or major depression (if not considered in remission)
* At risk of suicide in the opinion of the investigator
* Any abnormal MRI findings, such as presence of cerebral vascular pathology, cortical stroke, etc or inability to tolerate MRI procedures or contraindication to MRI
* Unstable or clinically significant cardiovascular (e.g., myocardial infarction), kidney or liver disease
* Uncontrolled hypertension
* Screening hemoglobin A1c (HbA1C) >8%
* Poor peripheral venous access
* History of cancer except:

If considered to be cured or If not being actively treated with anti-cancer therapy or radiotherapy

- Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (211):
- United States (48):
  - Imaging End Points Clinical Research, Scottsdale, Arizona
  - Health Initiatives Research, PLLC, Fayetteville, Arkansas
  - Clinical Trials Inc., Little Rock, Arkansas
  - Neuro-Therapeutics Inc., Pasadena, California
  - Desert Valley Medical Group, Rancho Mirage, California
  - Anderson Clinical Research, Inc., Redlands, California
  - University of California, Davis; Alzheimers Disease Center, Department of Neurology, Sacramento, California
  - UCSF - Memory and Aging Center, San Francisco, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - KI Health Partners, LLC; New England Institute for Clinical Research, Stamford, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - JEM Research LLC, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Renstar Medical Research, Ocala, Florida
  - Bioclinica Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Columbus Memory Center, Columbus, Georgia
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Alzheimers Disease Center; Neurology, Winchester, Massachusetts
  - Health Partners Institute for Education and Research, Saint Paul, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - University of Nebraska Medical Center; Dept of Neurological Sciences, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Summit, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Columbia University Medical Center, New York, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Behavioral Health Research, Charlotte, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - University of Cincinnati; Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - Ohio State University; College of Medicine, Columbus, Ohio
  - Dayton Center for Neuro Disorders, Dayton, Ohio
  - Summit Research Network Inc., Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Northeastern Pennsylvania Memory, Plains, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Neurology Clinic PC, Cordova, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - Gadolin Research, LLC, Beaumont, Texas
  - Texas Neurology PA, Dallas, Texas
  - Kerwin Research Center, LLC, Dallas, Texas
  - Alzheimers Disease & Memory Disorders Center; Department of Neurology Baylor College of Medicine, Houston, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
- Argentina (3):
  - Hospital Italiano, Buenos Aires
  - Universidad Maimonides, Caba
  - DAMIC, Córdoba
- Australia (4):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - Hornsby Ku-ring-gai Hospital; Division of Rehabilitation & Aged Care, Hornsby, New South Wales
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
- Belgium (3):
  - AZ Sint Jan, Bruges
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (6):
  - CCBR - Brasilia, Brasília, Federal District
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Centro Psiquiatria Sandra Ruschel Ltda, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Clínica Dr. Norton Sayeg LTDA - EPP, São Paulo, São Paulo
- Canada (12):
  - OCT Research ULC, Kelowna, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - True North Clinical Research-Halifax, Halifax, Nova Scotia
  - True North Clinical Research Kentville, Kentville, Nova Scotia
  - Providence Care; Mental Health Services, Kingston, Ontario
  - Parkwood Hospital; Geriatric Medicine, London, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - ALPHA Recherche Clinique, Québec
- China (2):
  - Beijing Union Hospital, Beijing
  - Tianjin Medical University General Hospital, Tianjin (天津)
- Denmark (2):
  - Aarhus Universitetshospital, Neurologisk Afdeling F, Demensklinikken, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
- Laane-Tallinna Keskhaigla, Tallinn, Estonia
- France (11):
  - Hopital Pellegrin; Cmrr Aquitaine, Bordeaux
  - Hôpital de Jour du Centre pour Personnes Âgées; Louis Pasteur Neurologie, Colmar
  - Hopital Roger Salengro; Service de Neurologie, Lille
  - CHU de Limoges Hopital Dupuytren; Service de Medecine Geriatrique, Limoges
  - Hopital Broca, Paris
  - CH Pitie Salpetriere; IM2A, Paris
  - Hôpital Maison Blanche, Reims
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHU de Rouen Hopital; Service de Neurologie, Rouen
  - Hop Guillaume Et Rene Laennec; Cmrr St Herblain, Saint-Herblain
  - Hopital des Charpennes, Villeurbanne
- Germany (7):
  - ECRC Experimental and Clinical Research Center, Charité Campus Berlin Buch, Memory Clinic, Berlin
  - Klinikum Joh.Wolfg.Goethe-UNI Zentrum d. Psychiatrie Klinik f. Psychiatrie Psychosomatik, Frankfurt
  - Universitätsklinikum Freiburg, Zentrum für Geriatrie und Gerontologie, Freiburg im Breisgau
  - Universitätsklinikum des Saarlandes Klinik f. Psychiatrie und Psychotherapie, Homburg/Saar
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Pharmakologisches Studienzentrum, Mittweida
  - Klinikum rechts der Isar der TU München; Klinik für Psychiatrie und Psychotherapie, München
- Israel (3):
  - Rambam Medical Center, Haifa
  - Sheba Medical Center; Psychiatry Department, Ramat Gan
  - Tel Aviv Sourasky Medical Center; Department of Neurology, Tel Aviv
- Italy (12):
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata; Neurologia, Rome, Lazio
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratell;Neurologia, Rome, Lazio
  - IRCCS "Centro S. Giovanni di Dio" Fatebenefratelli -UO Alzheimer, Brescia, Lombardy
  - Irccs Multimedica Santa Maria; Unita' Di Neurologia, Castellanza, Lombardy
  - IRCCS Ospedale San Raffaele; Centro Disturbi della Memoria, Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale Neurologico Besta; UO Neuropatologia, Milan, Lombardy
  - Ospedale S. Maria Nascente; Fondazione Don Gnocchi; Dip. Neurologia Riabilitativa, Milan, Lombardy
  - Ospedale Casati Passirana di Rho; Centro Regionale Alzheimer, Passirana, Lombardy
  - IRCCS Neuromed; Neurologia I-Centro studio e cura delle demenze e UVA, Pozzilli, Molise
  - AO Città della Salute e della Scienza Osp.S.Giov.Battista Molinette; SC Geriatria, Turin, Piedmont
  - A.O. Universitaria Pisana; Neurologia, Pisa, Tuscany
- Japan (22):
  - National Center for Geriatrics and Gerontology, Aichi
  - Inage Neurology and Memory Clinic, Chiba
  - Fukuoka Mirai Hospital, Fukuoka
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Tsukazaki Hospital, Hyōgo
  - Kagawa Prefectural Central Hospital, Kagawa
  - Fujisawa City Hospital, Kanagawa
  - National Hospital Organization Sagamihara National Hospital, Kanagawa
  - Ijinkai Takeda General Hospital, Kyoto
  - Rakuwakai Otowarehabilitation Hospital, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Nagano
  - Iwate Medical University Hospital, Numakunai
  - Katayama Medical Clinic, Okayama
  - Osaka University Hospital, Osaka
  - Asakayama General Hospital, Osaka
  - NHO Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka
  - Kanto Central Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Shinjuku Research Park Clinic, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
- Norway (2):
  - Akershus universitetssykehus HF; Nevroklinikken S203, Lørenskog
  - Oslo universitetssykehus HF Ullevål sykehus; Hukommelsesklinikken, Oslo
- Peru (2):
  - Clinica Internacional; Unidad De Investigacion, Lima
  - Hospital Nacional Dos de Mayo; Unidad de Investigacion de Neurologia, Lima
- Poland (4):
  - NZOZ Dom Sue Ryder, Bydgoszcz
  - Centrum Medyczne Euromedis Sp. z o.o., Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - NZOZ WCA, Wroclaw
- Portugal (4):
  - Hospital de Braga; Servico de Neurologia, Braga
  - HUC; Servico de Neurologia, Coimbra
  - Hospital Pedro Hispano; Servico de Neurologia, Matosinhos Municipality
  - Hospital Geral de Santo Antonio; Servico de Neurologia, Porto
- Russia (8):
  - LLC Baltic Medicine, Saint Petersburg, Sankt-Peterburg
  - State Healthcare Institution of Sverdlovsk Region Sverdlovsk Regional Clinical Psychiatric Hospita, Yekaterinburg, Sverdlovsk Oblast
  - State Autonomous Healthcare Institution "Republican Clinical Neurological Center, Kazan'
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan'
  - Institution of RAMS (Mental Health Research Center of RAMS), Moscow
  - City Clinical Psychiatry Hospital #1, Nizhny Novgorod
  - St Nicolas Psychiatric Hospital; Chair of Psychiatry and Narcology of St. Petersburg Medical Academy, Saint Petersburg
  - Nebbiolo Center for Clinical Trials, Tomsk
- Serbia (3):
  - Clinic for Mental disorders Dr Laza Lazarevic, Belgrade
  - Neurology clinic, Clinical Center of Serbia, Belgrade
  - Clinic for neurology, Clinical Center Kragujevac, Kragujevac
- Private Practice; the Osteoporosis Clinic, Johannesburg, South Africa
- South Korea (9):
  - Dong-A University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Borame Medical Center, Seoul
- Spain (21):
  - Hospital General Universitario de Elche; Servicio de Neurología, Elche, Alicante
  - Fundació ACE, BArcelon, Barcelona
  - Hospital General De Catalunya; Servicio de Neurologia, Sant Cugat del Vallès, Barcelona
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital Virgen del Puerto. Servicio de Neurología, Plasencia, Caceres
  - Hospital Universitario Marques de Valdecilla; Servicio de Neurología, Santander, Cantabria
  - Hospital la Magdalena; Servicio de Neurologia, Castellon, Castellon
  - Hospital Santa Caterina, Unitat de Valoració de la memoria i les demencies, Salt, Girona
  - Policlínica Guipuzkoa; Servicio de Neurología, Donosti-San Sebastián, Guipuzcoa
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Neurologia, Santiago de Compostela, LA Coruña
  - Hospital San Pedro; Servicio de Neurología, Logroño, La Rioja
  - Hospital Quiron de Madrid; Servicio de Neurologia, Pozuelo de Alarcón, Madrid
  - Clinica Universitaria de Navarra; Servicio de Neurología, Pamplona, Navarre
  - CAE Oroitu, Barakaldo, Vizcaya
  - Hospital Perpetuo Socorro, Servicio de Geriatria, Albacete
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitario de Burgos. Servicio de Neurología, Burgos
  - Hospital Universitario Reina Sofia; Servicio de Neurologia, Córdoba
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Complejo Asistencial Universitario de Salamanca; Servicio de Psiquiatría; CSM La Alamedilla, Salamanca
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
- Sweden (2):
  - Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo
  - Sahlgrenska Academy University,Neuroscience and Physiology;Departmt of Psychiatry and Neurochemistry, Mölndal
- Taiwan (5):
  - Changhua Christian Hospital; Neurology, Changhua County
  - Kaohsiung Medical University Hospital; Neurology, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital - Neurology, New Taipei City
  - National Taiwan University Hospital; Neurology, Taipei
  - Chang Gung Memorial Foundation - Linkou - Neurology, Taoyuan District
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty; Neurology, Ankara
  - Istanbul University Istanbul School of Medicine; Neurology, Istanbul
  - Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun
- United Kingdom (11):
  - The Fritchie Centre, Charlton Lane Centre, Charlon Lane, Leckhampton; The Fritchie Centre, Cheltenham
  - Surrey and Borders NHS Foundation Trust; Brain Science Research Unit, Chertsey
  - Sussex Partnership NHS Foundation Trust; Cognitive Treatment and Research unit, Crowborough
  - Ninewells Hospital, Dundee
  - NHS Lothian - Western General Hospital; NHS Lothian - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital; Clinical Research Facility, Glasgow
  - RE:Cognition Health, London
  - Charing Cross Hospital; Imperial Memory Unit, Level 10 West, London
  - Manchester Royal Infirmary, Manchester
  - John Radcliffe Hospital, Oxford
  - University Southampton NHS Foundation Trust; Wessex Neurologica Centre, Southampton

REFERENCES:
- [Derived] Hibar DP, Bauer A, Rabe C, Borlinghaus N, Jethwa A, Kollmorgen G, Di Domenico A, Zetterberg H, Blennow K, Masters CL, Sperling RA, Bittner T. Elecsys pTau217 plasma immunoassay detection of amyloid pathology in clinical cohorts. Alzheimers Dement. 2026 Jan;22(1):e71009. doi: 10.1002/alz.71009. PMID 41537338
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Teng E, Manser PT, Shah M, Pickthorn K, Hu N, Djakovic S, Swendsen H, Blendstrup M, Faccin G, Ostrowitzki S, Sink KM. The Use of Episodic Memory Tests for Screening in Clinical Trials for Early Alzheimer's Disease: A Comparison of the Free and Cued Selective Reminding Test (FCSRT) and the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). J Prev Alzheimers Dis. 2023;10(1):41-49. doi: 10.14283/jpad.2022.101. PMID 36641609
- [Derived] Ostrowitzki S, Bittner T, Sink KM, Mackey H, Rabe C, Honig LS, Cassetta E, Woodward M, Boada M, van Dyck CH, Grimmer T, Selkoe DJ, Schneider A, Blondeau K, Hu N, Quartino A, Clayton D, Dolton M, Dang Y, Ostaszewski B, Sanabria-Bohorquez SM, Rabbia M, Toth B, Eichenlaub U, Smith J, Honigberg LA, Doody RS. Evaluating the Safety and Efficacy of Crenezumab vs Placebo in Adults With Early Alzheimer Disease: Two Phase 3 Randomized Placebo-Controlled Trials. JAMA Neurol. 2022 Nov 1;79(11):1113-1121. doi: 10.1001/jamaneurol.2022.2909. PMID 36121669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 209 centers in 27 countries.
Pre-assignment Details: A total of 806 participants were enrolled at 209 centers. 4 participants did not receive any study treatment meaning that the modified intent-to-treat and safety populations consisted of 802 participants.
Period: Overall Study
Arm/Group | Placebo | Crenezumab
Started | 399 | 407
Completed | 0 | 0
Not Completed | 399 | 407
Not completed — Adverse Event | 9 | 6
Not completed — Death | 4 | 0
Not completed — Multiple Reasons | 1 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Study Terminated By Sponsor | 355 | 374
Not completed — Symptomatic Deterioration | 0 | 1
Not completed — Withdrawal by Subject | 28 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Crenezumab | Total
Number analyzed (Participants) | 399 | 407 | 806
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (7.9) | 71.1 (7.5) | 70.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 231 | 456
  Male | 174 | 176 | 350
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 42 | 35 | 77
  Not Hispanic or Latino | 334 | 348 | 682
  Not Stated | 15 | 19 | 34
  Unknown | 8 | 5 | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 8 | 5 | 13
  Asian | 45 | 47 | 92
  Black or African American | 4 | 3 | 7
  Multiple | 4 | 3 | 7
  Unknown | 5 | 7 | 12
  White | 333 | 342 | 675

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 77 in Clinical Dementia Rating-Sum of Boxes (CDR-SB) Scale Score
Description: The CDR-SB rates impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care) on a 5-point scale in which no impairment = 0, questionable impairment = 0.5 and mild, moderate and severe impairment = 1, 2 and 3 respectively. The score range is from 0 to 18 with a high score indicating a high disease severity. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline for this primary endpoint. Data after 29 January 2019 are censored for the primary and secondary efficacy analyses to avoid potential biases due to investigators, participants, raters, etc. being potentially influenced by early closure of the study due to lack of efficacy.
Time Frame: Baseline, Week 77
Population: The Modified Intent-To-Treat population (Placebo (n = 398); Cren (n = 404)) was defined as all randomized participants who received at least 1 dose of study drug, with participants grouped according to the treatment assigned at randomization. Data presented below is only for participants that were included in the actual analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | 3.19 (0.434) | 1.89 (0.471)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 1.30, 95% CI 2-sided [0.00 to 2.60], Standard Error of Mean 0.633

2. Secondary Outcome: Change From Baseline to Week 77 in Alzheimer's Disease Assessment Scale-Cognition 13 (ADAS-Cog-13) Subscale Score
Description: The ADAS-Cog-13 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Most of these are assessed by tests although some are rated by the clinician on a 5-point scale. The ADAS-Cog-13 is the ADAS-Cog-11 with 2 further items: delayed word recall and total digit cancellation. The score range for ADAS-Cog-13 is from 0 to 85 with high scores representing severe dysfunction. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | 8.90 (1.382) | 7.16 (1.526)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 1.74, 95% CI 2-sided [-2.40 to 5.89], Standard Error of Mean 2.028

3. Secondary Outcome: Change From Baseline to Week 77 in Alzheimer's Disease Assessment Scale-Cognition 11 (ADAS-Cog-11) Subscale Score
Description: The ADAS-Cog-11 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Most of these are assessed by tests although some are rated by the clinician on a 5-point scale. The score range for ADAS-Cog-11 is from 0 to 70 with high scores representing severe dysfunction. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | 7.16 (1.452) | 6.84 (1.592)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.33, 95% CI 2-sided [-4.03 to 4.68], Standard Error of Mean 2.124

4. Secondary Outcome: Change From Baseline to Week 77 on Severity of Dementia, Assessed Using the CDR-Global Score (CDR-GS)
Description: The CDR-GS represents a semi-structured interview which rates impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care) on a 5-point scale in which CDR 0 = no dementia and CDR 0.5, 1, 2 or 3 = questionable, mild, moderate or severe dementia respectively. The range in scores for the CDR-GS is from 0 to 3 and a high score on the CDR-GS would indicate a high disease severity. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | 0.39 (0.096) | 0.29 (0.102)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.09, 95% CI 2-sided [-0.20 to 0.39], Standard Error of Mean 0.141

5. Secondary Outcome: Change From Baseline to Week 77 on Severity of Dementia, Assessed Using the Mini Mental State Evaluation (MMSE)
Description: The MMSE is a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target 6 areas: orientation, registration, attention, short-term recall, language and constructional praxis/visuospatial abilities. The scores on the MMSE range from 0 to 30, with higher scores indicating better function. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | -3.63 (0.672) | -3.21 (0.740)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.41, 95% CI 2-sided [-2.42 to 1.60], Standard Error of Mean 0.985

6. Secondary Outcome: Change From Baseline to Week 77 on Function as Assessed by (ADCS-ADL) Total Score
Description: The ADCS-ADL (Alzheimer's Disease Cooperative Study-Activities of Daily Living) is the scale most widely used to assess functional outcomes in participants with AD. The ADCS-ADL covers both basic ADL (e.g., eating and toileting) and more complex 'instrumental' ADL or iADL (e.g., using the telephone, managing finances and preparing a meal). The ADCS-ADL consists of 23 questions with a score range of 0 to 78 where a higher score represents better function. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | -8.83 (2.064) | -6.31 (2.278)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -2.52, 95% CI 2-sided [-8.74 to 3.70], Standard Error of Mean 3.052

7. Secondary Outcome: Change From Baseline to Week 77 on Function as Assessed by (ADCS-iADL) Instrumental Score
Description: The ADCS-iADL (Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living) measures activities such as using the telephone, managing finances and preparing a meal. The ADCS-iADL consists of 16 questions with a score range of 0 to 56 where a higher score represents better function. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | -6.69 (1.692) | -5.51 (1.872)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -1.19, 95% CI 2-sided [-6.29 to 3.92], Standard Error of Mean 2.501

8. Secondary Outcome: Change From Baseline to Week 77 on Function as Assessed by the Functional Activities Questionnaire (FAQ) Total Score
Description: The Functional Activities Questionnaire (FAQ) is an instrument consisting of 10 items and assesses instrumental, social and cognitive functioning. The score range is from 0 to 30 with higher scores representing higher impairment. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | 5.00 (0.991) | 4.37 (1.059)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 0.63, 95% CI 2-sided [-2.25 to 3.51], Standard Error of Mean 1.420

9. Secondary Outcome: Change From Baseline to Week 77 on a Measure of Dependence Level Assessed From the ADCS-ADL Score
Description: as for outcome 6
Time Frame: Baseline, Week 77
Population: Please note that for this Outcome Measure, no participants were evaluated at all as the derivation of this endpoint was not pre-specified before the Sponsor terminated the study and therefore it was not reported.
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline to Week 53 on Behavior in Neuropsychiatric Inventory Questionnaire (NPI-Q) Total Score
Description: The NPI-Q evaluates 12 neuropsychiatric disturbances common in dementia: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavioral disturbances and appetite/eating abnormalities. The severity of each neuropsychiatric symptom is rated on a 3-point scale (mild, moderate and marked). The total severity score range is from 0 to 36 with higher scores representing higher severity. Difference in mean change from Baseline to Week 53 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures adjusting for disease severity, APOEe4 status, geographic region and the use/non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 53
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 102 | 110
Units on a Scale | -0.00 (0.852) | 0.76 (0.886)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.76, 95% CI 2-sided [-1.75 to 0.23], Standard Error of Mean 0.502

11. Secondary Outcome: Quality of Life-Alzheimer's Disease (QoL-AD) Scale Score
Description: The QoL-AD (Quality of Life - Alzheimer's Disease) scale assesses QoL in participants who have dementia. The QoL-AD consists of 13 items covering aspects of participants' relationships with friends and family, physical condition, mood, concerns about finances and overall assessment of QoL. Items are rated on 4-point Likert-type scales ranging from 1 [poor] to 4 [excellent]. The score range is from 13 to 52, with higher scores indicating a better QoL. The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 11
Units on a Scale | -1.61 (1.310) | -1.16 (1.432)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.46, 95% CI 2-sided [-3.30 to 2.39], Standard Error of Mean 1.383

12. Secondary Outcome: Zarit Caregiver Interview for Alzheimer's Disease (ZCI-AD) Scale Score
Description: The ZCI-AD is a modified version of the Zarit Burden Interview, which was originally designed to reflect the stresses experienced by caregivers of people with dementia. This modified version includes slight modifications in item and title wording (e.g., removal of "your relative" to refer directly to the patient, removal of "burden" from title) and the use of 11-point numerical rating scales. The ZCI-AD scale consists of a total of 30 items. Total scores will be calculated with a total score range from 0 to 300 (higher scores indicate a higher burden on the caregiver). The difference in mean change from Baseline to Week 53 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 53
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 101 | 108
Units on a Scale | 9.20 (9.292) | 2.65 (9.643)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 6.55, 95% CI 2-sided [-4.35 to 17.44], Standard Error of Mean 5.527

13. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Questionnaire Domain Scores for Participants
Description: The EQ-5D is a standardized measure of health status designed to provide a simple generic measure of health for clinical and economic appraisal. It is broadly applicable across a wide range of health conditions and treatment. The EQ-5D assesses five domains to provide a health state index. These are anxiety/depression, pain/discomfort, usual activities, mobility, and self-care. The scores on the EQ-5D ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). The difference in mean change from Baseline to Week 77 between Crenezumab and Placebo treated participants was estimated. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | -3.69 (3.961) | -3.39 (4.392)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-12.31 to 11.71], Standard Error of Mean 5.831

14. Secondary Outcome: European Quality of Life-5 Dimensions (EQ-5D) Questionnaire Domain Scores for Caregivers
Description: as for outcome 13
Time Frame: Baseline, Week 77
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 15 | 12
Units on a Scale | -4.07 (2.724) | -0.68 (3.031)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -3.38, 95% CI 2-sided [-11.50 to 4.73], Standard Error of Mean 3.940

15. Secondary Outcome: Percentage of Participants With Adverse Event (AEs) and Serious Adverse Event (SAEs)
Description: An Adverse Event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up until 16 weeks after the last dose of study drug (up to 117 weeks).
Population: The Safety analysis population included all randomized participants who received at least 1 dose of study drug with participants grouped according to actual treatment received. If a participant received at least 2 vials of crenezumab, then they were placed in the crenezumab arm.
Measure: Number; unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 398 | 404
Percentage
  AEs | 73.1 | 73.5
  SAEs | 10.6 | 8.2

16. Secondary Outcome: Percentage of Participants With Anti-Crenezumab Antibodies
Description: Participants were considered positive or negative for ADA based on their baseline and post-baseline sample results. The number and percentage of participants with confirmed positive ADA levels were determined for Crenezumab and Placebo groups. The prevalence of ADA at baseline was calculated as the proportion of participants with confirmed positive ADA levels at baseline relative to the total number of participants with a sample available at baseline. The incidence of treatment-emergent ADAs was determined as the proportion of participants with confirmed post-baseline positive ADAs relative to the total number of participants that had at least one post-baseline sample available for ADA analysis.
Time Frame: Baseline up to Week 105
Population: Please note that for this Outcome Measure, no Participants were evaluated at all as the existing immunogenicity data from an identical study (Study BN29552) showed a low potential of Crenezumab to induce Anti-Drug Antibodies (ADAs).
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Serum Concentration of Crenezumab
Description: Serum concentration data for Crenezumab will be tabulated and summarized. Descriptive summary statistics will include the arithmetic mean and SD. Since a sparse PK sampling design is being used, population (non-linear mixed-effects) modeling will be used to analyze the dose concentration-time data of crenezumab. Information from other clinical studies may be incorporated to establish the PK model. Please note that Post-dose samples were not collected at Weeks 5, 13, 37, 53 and 77.
Time Frame: Pre-infusion (0 hour), 60-90 minutes post-infusion on Day 1 Week 1 and on Week 25; Weeks 13 (Pre-dose), 37 (Pre-dose), 53 (Pre-dose) and 77 (Pre-dose) (infusion length = as per the Pharmacy Manual)
Population: The PK Analysis population was defined as all participants who have received at least one dose of crenezumab and with at least one evaluable post-dose PK sample. Data presented below is only for participants that were included in the actual analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Crenezumab
Number analyzed (Participants) | 138
ug/mL
  Week 1 Day 1 Predose | NA (NA) — No Drug was administered at this point so no concentrations detected.
  Week 1 Day 1 Postdose: number analyzed (Participants) | 110
  Week 1 Day 1 Postdose | 1260 (437)
  Week 5 Predose | 246 (128)
  Week 13 Predose: number analyzed (Participants) | 128
  Week 13 Predose | 360 (162)
  Week 25 Predose: number analyzed (Participants) | 125
  Week 25 Predose | 401 (196)
  Week 25 Postdose: number analyzed (Participants) | 106
  Week 25 Postdose | 1650 (443)
  Week 37 Predose: number analyzed (Participants) | 97
  Week 37 Predose | 456 (351)
  Week 53 Predose: number analyzed (Participants) | 32
  Week 53 Predose | 401 (130)
  Week 77 Predose: number analyzed (Participants) | 3
  Week 77 Predose | 357 (94.2)

18. Secondary Outcome: Plasma Amyloid Beta (Abeta) 40 Concentrations
Description: Plasma Abeta 40 concentrations will be measured over time and descriptive summary statistics will include the arithmetic mean and SD. Please note that Pre-dose samples were only collected at Weeks 1 and 53.
Time Frame: Week 1 Day 1; Weeks 53
Population: The PD Analysis population was defined as all participants who have received at least one dose of crenezumab and with at least one evaluable post-dose PK sample. Data presented below is only for participants that were included in the actual analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crenezumab
Number analyzed (Participants) | 36
ng/mL
  Week 1 Day 1 Predose | 0.415 (0.0687)
  Week 53 Predose: number analyzed (Participants) | 13
  Week 53 Predose | 46.6 (6.91)

19. Secondary Outcome: Plasma Amyloid Beta (Abeta) 42 Concentrations
Description: Plasma Abeta 42 concentrations will be measured over time and descriptive summary statistics will include the arithmetic mean and SD. Please note that Pre-dose samples were only collected at Weeks 1 and 53.
Time Frame: Week 1 Day 1; Weeks 53
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crenezumab
Number analyzed (Participants) | 36
ng/mL
  Week 1 Day 1 Predose | 0.0331 (0.00463)
  Week 53 Predose: number analyzed (Participants) | 13
  Week 53 Predose | 2.94 (0.473)

20. Secondary Outcome: Percentage Change From Baseline to Week 105 in Whole Brain Volume as Determined by Magnetic Resonance Imaging (MRI)
Description: Percentage Change in Whole Brain Volume will be measured over time and descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 4 | 4
Percentage | -2.71 (0.444) | -2.15 (0.345)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.56, 95% CI 2-sided [-2.01 to 0.89], Standard Error of Mean 0.622

21. Secondary Outcome: Percentage Change From Baseline to Week 105 in Ventricle Volume as Determined by Magnetic Resonance Imaging (MRI)
Description: Percentage Change in Ventricle Volume will be measured over time and descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 4 | 4
Percentage | 18.78 (1.343) | 17.18 (1.145)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = 1.60, 95% CI 2-sided [-1.70 to 4.90], Standard Error of Mean 1.668

22. Secondary Outcome: Percentage Change From Baseline to Week 105 in Hippocampal Volume as Determined by Magnetic Resonance Imaging (MRI)
Description: Percentage Change in Hippocampal Volume will be measured over time and descriptive summary statistics will include the arithmetic mean, median, range, SD, and coefficient of variation, as appropriate. Mixed model repeated measures (MMRMs) adjusting for disease severity, APOEe4 status, geographic region, and the use or non-use of anti-dementia medications at baseline were used to estimate the mean change from baseline.
Time Frame: Baseline, Week 105
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Crenezumab
Number analyzed (Participants) | 2 | 2
Percentage | -6.34 (0.338) | -5.98 (0.290)
Statistical Analysis 1: Comparison: Placebo vs Crenezumab; Test type: Superiority; Least Squares Mean Difference = -0.36, 95% CI 2-sided [-1.13 to 0.41], Standard Error of Mean 0.373

ADVERSE EVENTS:
Time Frame: Baseline up until 16 weeks after the last dose of study drug (up to 117 weeks).
Arm/Group | Placebo | Crenezumab
All-Cause Mortality (participants affected / at risk) | 6/398 | 0/404
Serious Adverse Events (participants affected / at risk) | 42/398 | 33/404
Other Adverse Events (participants affected / at risk) | 77/398 | 85/404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=398) | Crenezumab (N=404)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
TRIFASCICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0)
SUDDEN DEATH (General disorders) | 2 (2) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 1 (1)
ENTEROBACTER PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
NEUROSYPHILIS (Infections and infestations) | 0 (0) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
ARTHROSCOPY (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE GIANT CELL TUMOUR MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CLEAR CELL ENDOMETRIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL ARTERIOSCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
SPEECH DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
SUPERIOR SAGITTAL SINUS THROMBOSIS (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 2 (2) | 0 (0)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
DELUSION (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDE THREAT (Psychiatric disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CARDIAC ABLATION (Surgical and medical procedures) | 0 (0) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=398) | Crenezumab (N=404)
NASOPHARYNGITIS (Infections and infestations) | 25 (32) | 24 (28)
FALL (Injury, poisoning and procedural complications) | 20 (34) | 19 (26)
HEADACHE (Nervous system disorders) | 22 (28) | 25 (30)
HYPERTENSION (Vascular disorders) | 15 (18) | 27 (29)

LIMITATIONS AND CAVEATS:
This study was discontinued due to an interim analysis in the BN29552 study, which indicated that Crenezumab was unlikely to meet its primary endpoint. No participants reached Week 105 for primary and secondary efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT03114657/Prot_SAP_000.pdf